CLINICAL TRIAL: NCT04669756
Title: Ovariopexy for Adhesion Prevention After Laparoscopic Removal of Endometriosis of the Pelvic Side Wall or the Ovary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. med. Sebastian Daniel Schäfer, Head of Gynecology, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Schäfer_Endo_Ovariopexie
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Endometriosis; Adhesion; Surgery
Keywords: endometriosis; ovariopexy; adhesion prevention; laparoscopy; complications; AMH
MeSH Terms: conditions — Endometriosis; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Experimental): ovariopexy for 2 days
  Interventions: Procedure: ovariopexy
- B (Experimental): ovariopexy for 4 days
  Interventions: Procedure: ovariopexy
- C (Experimental): ovariopexy for 6 days
  Interventions: Procedure: ovariopexy
- D (Placebo Comparator): Placebo Operation for 2 days
  Interventions: Procedure: placebo operation

INTERVENTIONS:
Procedure: ovariopexy — if endometriosis was removed from the pelvic side wall or the ovary or both leading to an open wound adjacent to the ovary, ovariopexy was performed on both sides using a transabdominal-transovarian suture being tied extracorporeally on the patients Skin leading to uplifting of the ovary to the abdominal wall
  Arms: A; B; C
Procedure: placebo operation — in arm D sutures are transabdominal only
  Arms: D

SUMMARY:
prospective randomized Trial comparing ovariopexy over 2, 4 or 6 days vs Placebo after surgery because of endometriosis of the pelvic side wall or the ovary or both

ELIGIBILITY:
Inclusion Criteria:

* premenopausal
* wants to participate
* removal of endometriosis of the pelvic side wall or ovary

Exclusion Criteria:

* postmenopausal
* cannot give informed consent
* no endometriosis during Operation
* no Opening of pelvic side wall or ovary during the Operation
* pregnant
* breast feeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 409 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
prevalence of postoperative ovarian adhesions | 3 months after operation
  prevalence of postoperative ovarian adhesions

SECONDARY OUTCOMES:
postoperative pain | daily during postoperative hospitalisation and at follow up visit after 3 months
  postoperative pain (NRS)
AMH | at follow up visit after 3 months
  AMH level
postoperative infectious complications | up to 3 months after operation
  postoperative infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian D Schaefer, MD PhD, Principal Investigator — University Hospital Muenster, Germany
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
data can be shared upon reasonable request and according to regulations